CLINICAL TRIAL: NCT02054598
Title: The CHOICES/OPCIONES Project: Improving Colon Cancer Screening for Diverse Populations
Brief Title: Improving Colon Cancer Screening for Diverse Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of New Mexico (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 09-0537
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Usual care.
- Intervention group (Experimental): Decision aid and navigation
  Interventions: Behavioral: Decision aid and navigation

INTERVENTIONS:
Behavioral: Decision aid and navigation — Patients in the intervention group will receive a combined intervention consisting of a CRC screening decision aid and assistance from a trained patient navigator.
  Arms: Intervention group

SUMMARY:
This study is a multi-site randomized, controlled trial testing the effect of a combined intervention that includes a colorectal cancer (CRC) screening decision aid plus patient navigation in a diverse, primary care patient population in clinical sites in North Carolina and New Mexico.

Our primary aim is to determine the effect of the intervention on CRC screening completion six months after the index visit among all enrolled participants and among Latinos. Secondarily, we will determine how this intervention affects screening-related knowledge, self-efficacy, intent, and clinical communication, and examine whether these factors mediate the effect of the intervention on screening test completion. Lastly, we will explore whether insurance status, ethnicity, and patient language preference moderate the effect of the intervention on screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 to 75 years old who are not current with colorectal cancer (CRC) screening, defined as not having completed a home fecal occult blood test (FOBT) within the past year; a flexible sigmoidoscopy within the past five years; or a colonoscopy within the past ten years.
* Have an appointment at one of the clinic sites

Exclusion Criteria:

* Will include: inability to speak either English or Spanish, severe illness at the time of the clinic visit, co-morbidity that is estimated to limit life-expectancy to less than 5 years as estimated by the treating nurse or provider, severe cognitive, visual, or hearing impairment that would preclude Decision Aid (DA) viewing. We will also exclude patients who are at elevated risk for CRC, defined as having ever been diagnosed with CRC, a precancerous (adenomatous) polyp, or inflammatory bowel disease.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening completion | 6 months
  A blinded medical record review will be used to determine the primary outcome of 6 month Colorectal cancer screening status. To ensure optimal capturing of screening test completion, we will ask participants whose medical record does not contain evidence of screening to verify non-completion during the 6 month phone survey.

SECONDARY OUTCOMES:
Colorectal cancer screening knowledge | Post-encounter measure
  Following the provider encounter, we will administer the post-encounter survey to measure intermediate screening related knowledge.
Colorectal cancer screening related self-efficacy | 6 months
  The Colorectal cancer screening self-efficacy will be measured by the post-encounter survey.
Colorectal cancer screening related intent | 6 months
  The post-encounter survey will be used to measure the Colorectal cancer screening related intent.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Reuland, MD, MPH, Principal Investigator — University of North Carolina
Locations (3):
- United States (3):
  - University of New Mexico, Albuquerque, New Mexico
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Healthcare Systems, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reuland DS, Brenner AT, Hoffman R, McWilliams A, Rhyne RL, Getrich C, Tapp H, Weaver MA, Callan D, Cubillos L, Urquieta de Hernandez B, Pignone MP. Effect of Combined Patient Decision Aid and Patient Navigation vs Usual Care for Colorectal Cancer Screening in a Vulnerable Patient Population: A Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):967-974. doi: 10.1001/jamainternmed.2017.1294. PMID 28505217
- [Derived] Brenner AT, Hoffman R, McWilliams A, Pignone MP, Rhyne RL, Tapp H, Weaver MA, Callan D, de Hernandez BU, Harbi K, Reuland DS. Colorectal Cancer Screening in Vulnerable Patients: Promoting Informed and Shared Decisions. Am J Prev Med. 2016 Oct;51(4):454-62. doi: 10.1016/j.amepre.2016.03.025. Epub 2016 May 27. PMID 27242081
- [Derived] Brenner AT, Getrich CM, Pignone M, Rhyne RL, Hoffman RM, McWilliams A, de Hernandez BU, Weaver MA, Tapp H, Harbi K, Reuland D. Comparing the effect of a decision aid plus patient navigation with usual care on colorectal cancer screening completion in vulnerable populations: study protocol for a randomized controlled trial. Trials. 2014 Jul 8;15:275. doi: 10.1186/1745-6215-15-275. PMID 25004983